CLINICAL TRIAL: NCT02190565
Title: Supplementation With WellnessPack Mama During Pregnancy and Lactation - a Randomized Double-blind, Placebo-controlled Study
Brief Title: Safety and Efficacy Study of a Food Supplement for Pregnant and Lactating Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision - strategy changes and budget limitations
Sponsor: Oriflame Cosmetics AB (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014/815-31/4
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Anaemia
Keywords: pregnancy, lactation, food supplement, anaemia
MeSH Terms: conditions — Anemia; Breast Feeding | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo consisting of two sham multivitamin and mineral tablets and two capsules of oil
  Interventions: Dietary Supplement: Food supplement
- Food supplement (Active Comparator): Food supplement consisting of fish oil (omega 3 fatty acids DHA and EPA) and multivitamin and mineral tablets with extra iron and folic acid
  Interventions: Dietary Supplement: Food supplement

INTERVENTIONS:
Dietary Supplement: Food supplement — Randomized double-blind, placebo-controlled
  Other Names: WellnessPack mama

SUMMARY:
The purpose of this study is to determine whether a food supplement consisting of vitamins, minerals and fish oil taken during and after pregnancy can decrease the need for additional iron supplementation due to anemia during pregnancy, and optimize levels of nutritional markers such as vitamin D and docosahexaenoic acid (DHA, an omega 3 fatty acid) in maternal blood and breast milk, compared to placebo.

DETAILED DESCRIPTION:
200 healthy, pregnant women will be randomized to receive either active or placebo at their first visit to the pre-natal centres. They will be monitored at regular intervals, blood samples will be taken and they will be asked about compliance and any adverse reactions.

Approx 8 weeks after delivery, the women will come to the pre-natal centres for a check-up. During this visit, a blood sample will be drawn and a breast milk sample will be collected.

The blood samples will be analysed for haemoglobin, serum ferritin, vitamin D and DHA. The breast milk samples will be analysed for vitamin D and DHA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women aged 18-40 years with a body mass index (BMI) above 18.5 and below 35 kg/m2 who visit pre-natal clinics (midwife centres) to register.
* Nulliparous and multiparous women.
* The women must be able to understand verbal and written information in Swedish to give an informed consent to participate in the study.

Exclusion Criteria:

* Women below the age of 18 or above 40 years old.
* Women with a BMI below 18.5 or above 35 kg/m2.
* Women with any form of anaemia as diagnosed at the first visit to the prenatal clinic.
* Women expecting two or more babies.
* Women who have undergone bariatric surgery.
* Women on medication with pharmaceuticals that could affect the result of the study, e.g., vitamin K antagonists.
* Women who are allergic to any of the components of WellnessPack mama, e.g., fish.
* Women who suffer from drug or alcohol abuse.
* Women who suffer from known severe eating disorders.
* Women who suffer from chronic diseases that could affect gastrointestinal absorption and metabolism.
* Women who want to continue or start using similar food supplements in addition to WellnessPack mama/placebo, unless recommended by a physician or midwife, will be excluded from the study.
* Upon miscarriage or transfer to prenatal care specialist, the subject is excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-04-07 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of anaemia in active and placebo groups | pregnancy week 28-30
  Blood will be analysed for haemoglobin and ferritin values. We will compare how many women in each group (active vs placebo) are ordinated iron supplementation due to anaemia by mid-pregnancy.

SECONDARY OUTCOMES:
Levels of nutritional biomarkers in maternal blood and breast milk | 6-10 weeks after delivery
  Levels of nutritional biomarkers such as DHA and vitamin D in maternal blood and breast milk will be measured in active and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Lindén Hirschberg, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Woman and Child Health, Division of Obstetrics and Gynecology, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Background] Kawai K, Spiegelman D, Shankar AH, Fawzi WW. Maternal multiple micronutrient supplementation and pregnancy outcomes in developing countries: meta-analysis and meta-regression. Bull World Health Organ. 2011 Jun 1;89(6):402-411B. doi: 10.2471/BLT.10.083758. Epub 2011 Mar 21. PMID 21673856
- See also: World Health Organization. Worldwide prevalence of anaemia 1993-2005: WHO Global Database on Anaemia. — http://whqlibdoc.who.int/publications/2008/9789241596657_eng.pdf